CLINICAL TRIAL: NCT03487094
Title: Growth Monitoring Study of Infants Fed Formula for 16 Weeks
Brief Title: Growth and Tolerance of Infants Fed Formula for 16 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nature's One (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: N1.2018
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Child Development
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: Multi-Investigator, Prospective, Randomized Clinical Trial
Masking Description: Eligible infants are randomized to commercial control or experimental product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Growth, Tolerance of Infants-Exp (Active Comparator): Infant Formula
  Interventions: Other: Infant formula
- Growth,Tolerance of Infants-Com (Active Comparator): Infant Formula
  Interventions: Other: Infant formula

INTERVENTIONS:
Other: Infant formula — Multi-centered, prospective, randomized clinical trial

SUMMARY:
Growth and Tolerance Trial of Iron-fortified infant formulas

DETAILED DESCRIPTION:
16 WEEK GROWTH AND TOLERANCE

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants, 37-42 weeks gestational age

Exclusion Criteria:

* Any condition that would negatively impact assessment of growth and tolerance

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 216 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Growth | 16 weeks
  Weight Gain

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Murray, MD, Study Director — Consultant
Locations (24):
- United States (24):
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Harris Pediatric Clinic, Newport, Arkansas
  - Searcy Medical Center, Searcy, Arkansas
  - Norwich Pediatric Group, PC, Norwich, Connecticut
  - Pediatrics by the Sea, Delray Beach, Florida
  - Altamonte Pediatric Associates, Lake Mary, Florida
  - New Horizon Research Center, Miami, Florida
  - Paramount Research Solutions, College Park, Georgia
  - Qualmedica Research, Evansville, Indiana
  - Qualmedica Research, Owensboro, Kentucky
  - Portico Pediatrics, Shreveport, Louisiana
  - Gvozden Pediatrics, Millersville, Maryland
  - Valley Stream Pediatrics_Lashley, Valley Stream, New York
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Pediatric Partners, Raleigh, North Carolina
  - Piedmont Healthcare, Statesville, North Carolina
  - Aventiv Research, Inc, Columbus, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Cynthia Strieter-Boland, MD, Westlake, Ohio
  - Red Lion Pediatrics, Bensalem, Pennsylvania
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Coastal Pediatric Research, North Charleston, South Carolina
  - Southwestern Children's Research Associates, PA, San Antonio, Texas
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia